CLINICAL TRIAL: NCT07273747
Title: A Randomized Controlled Trial on the Effects of Oral Kelulut Honey Supplementation on Conjunctival Goblet Cell Density, Tear Film Stability, Dry Eye Disease Symptoms and Vision-Related Function in Patients With Allergic Conjunctivitis
Brief Title: Kelulut Honey for Allergic Conjunctivitis and Dry Eye Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shahidatul Adha Mohamad, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/KK/24080659
Record Dates: First submitted 2025-11-28; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Symptoms; Allergic Conjunctivitis of Both Eyes
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kelulut Honey 60 g (KH-60) (Experimental): Kelulut honey is provided in pre-packaged 30 g sachets to standardize dosing and maintain blinding across study arms.
  Interventions: Dietary Supplement: Kelulut Honey 60 g Oral Supplement
- Kelulut Honey 120 g (KH-120) (Experimental): Kelulut honey is provided in pre-packaged 30 g sachets to standardize dosing and maintain blinding across study arms.
  Interventions: Dietary Supplement: Kelulut Honey 120 g Oral Supplement
- Placebo (Placebo Comparator): The placebo consists of a honey-flavoured zero-calorie syrup, pre-packaged in sachets identical to the Kelulut honey sachets to maintain blinding.
  Interventions: Other: Honey-Flavoured Zero-Calorie Syrup (Placebo)

INTERVENTIONS:
Dietary Supplement: Kelulut Honey 60 g Oral Supplement — Participants in this arm will consume two 30 g sachets of Kelulut honey once daily (total 60 g/day) for one month. The honey will be taken directly from the sachet without dilution, on an empty stomach, 30 minutes before breakfast. Participants will continue their usual treatment for allergic conjunctivitis and dry eye disease.
  Other Names: KH-60; Group A
  Arms: Kelulut Honey 60 g (KH-60)
Dietary Supplement: Kelulut Honey 120 g Oral Supplement — Participants in this arm will consume four 30 g sachets of Kelulut honey daily (total 120 g/day) for one month. The daily dose will be divided into two administrations: two sachets before breakfast or lunch, and two sachets before dinner. The honey will be taken directly from the sachets without dilution, at least 30 minutes before meals. Participants will continue their usual treatment for allergic conjunctivitis and dry eye disease.
  Other Names: KH-120; Group B
  Arms: Kelulut Honey 120 g (KH-120)
Other: Honey-Flavoured Zero-Calorie Syrup (Placebo) — Participants in this placebo group will receive honey-flavoured zero-calorie syrup, pre-packaged in sachets identical to those used for the Kelulut honey. Each participant will consume two sachets per day, to be taken daily, once before breakfast, for one month duration. The syrup is to be taken directly from the sachets, without dilution, before meals.
  Other Names: Group C; KH-P
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if oral Kelulut honey works to improve eye symptoms in adults with allergic conjunctivitis. It will also look at how safe Kelulut honey is when taken as a daily supplement.

The main questions it aims to answer are:

1. Does oral Kelulut honey reduce itchy, red, watery eyes and dry eye symptoms in people with allergic conjunctivitis?
2. Does oral Kelulut honey improve tear film stability and the health of conjunctival goblet cells (special cells on the eye surface that help keep the eye moist)?
3. What side effects or medical problems do participants have when taking Kelulut honey?

Researchers will compare oral Kelulut honey to a honey-flavoured placebo syrup (a look-alike drink that does not contain Kelulut honey) to see if Kelulut honey is more effective than placebo for treating eye symptoms in allergic conjunctivitis.

Participants will:

1. Take either oral Kelulut honey or a honey-flavoured placebo syrup every day for 1 month
2. Continue their usual treatment for allergic conjunctivitis and dry eye disease as prescribed by their eye doctor
3. Attend clinic visits for eye check-ups, including tests of tear film stability, dry eye symptoms, and eye surface health
4. Answer questionnaires about their eye symptoms and how these affect their daily activities and vision-related quality of life

Participation is voluntary, and participants may stop taking part in the study at any time. Data collected up to the time they withdraw may still be used for research, but their routine medical care will not be affected

ELIGIBILITY:
Inclusion Criteria:

i. Age between 18-40 years old ii. Confirmed diagnosis of allergic conjunctivits iii. Ocular surface disease index (OSDI) score > 12 iv. Compliance to conventional allergic conjunctivitis treatment

Exclusion Criteria:

i. Any corneal or ocular surface pathology ii. Known diabetes mellitus or impaired glucose test iii. Ocular surface disease due to trachoma or other inflammatory conditions iv. Consume anti-inflammatory medications such as steroids, NSAIDS, oral doxycycline v. Concurrent use of other supplements or alternative therapies such as royal jelly, Manuka honey eye drop or omega-3 fatty acid vi. Using preservative-containing topical eye drops for ocular problems other than AC, such as anti-glaucoma medication vii. History of ocular trauma/surgery or refractive surgery within last 3 years viii. Wearing contact lens in the last 3 months ix. Underlying inflammatory/ systemic disease and connective tissue diseases x. Recent conjunctivitis in the last 3 months xi. Patients on immunosuppressant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in conjunctival goblet cell density (GCD) | Baseline and 1 month
  Goblet cell density measured via impression cytology and quantified using standard morphological grading. Change from baseline to 1 month will be compared between groups.

SECONDARY OUTCOMES:
Change in tear film break-up time (TBUT) | Baseline and 1 month
  TBUT measured using fluorescein dye under slit-lamp examination. Change from baseline to 1 month will be compared between groups.
Change in ocular surface staining score (OGS) | Baseline and 1 month
  Corneal and conjunctival fluorescein staining graded using the Oxford Grading Scheme (0-5). Change from baseline to 1 month will be compared between groups.
Change in Ocular Surface Disease Index (OSDI) score | Baseline and 1 month
  OSDI questionnaire score assessing dry eye symptoms and functional impact. Change from baseline to 1 month will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shahidatul Adha Dr, MD, MMed, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study is single-center, involves a small sample size, and institutional data governance policies do not permit open sharing of identifiable clinical data.